CLINICAL TRIAL: NCT05556590
Title: Impact of Preoperative Quantitative Flow Ratio on Radial Artery Graft Outcome After Coronary Artery Bypass Grafting in the ASRAB-Pilot Trial
Brief Title: Quantitative Flow Ratio on Radial Artery Graft Outcome After Coronary Artery Bypass Grafting
Acronym: ASRAB-QUARGO
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and director, Department of Cardiac Surgery,Vice President of Ruijin Hospital, Ruijin Hospital
Other Study IDs: KY-2022144
Record Dates: First submitted 2022-09-06; First posted 2022-09-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass grafting; Radial artery graft; Quantitative flow ratio
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- QFR-Low Group: Based on preoperative CAG, QFR analysis will be conducted for vessels bypassed with RA grafts. The RA-grafted vessels with QFR below the best cut-off value (0.50-0.55 assumed) will be allocated to QFR-Low group.
- QFR-High Group: Based on preoperative CAG, QFR analysis will be conducted for vessels bypassed with RA grafts. The RA-grafted vessels with QFR over the best cut-off value (0.50-0.55 assumed) will be allocated to QFR-High group.

SUMMARY:
In coronary artery bypass grafting (CABG), the use of radial artery (RA) is recommended by the guidelines only to significantly stenosed vessel, due to its high vulnerability to competitive flow. Fractional flow reserve (FFR) is the gold standard to measure physiological significance of coronary lesions and the potential for competitive flow. This study aims to investigate whether the preoperative quantitative flow ratio (QFR) measurement, a novel coronary angiography-based FFR, is associated with RA graft failure post-CABG, and to explore the best cut-off value of QFR for RA grafts using.

Patients from ASRAB-pilot trial (NCT04310995) undergoing primary isolated CABG using RA grafts, and with preoperative coronary angiography (CAG) images available for QFR analysis will be enrolled in this prospective double-blind observational study. QFR analysis will be conducted for all RA-grafted vessels based on preoperative CAG. The primary outcome will RA graft failure (FitzGibbon Grade B,O or S) evaluated by coronary computer tomography angiography or CAG at 7 days and 6 months post-CABG.

DETAILED DESCRIPTION:
Introduction:

The radial artery (RA) was first used by Carpentier for coronary artery bypass grafting (CABG) in 1971 because of a number of potential advantages, including ease of harvesting, a low propensity for wound infection, a larger diameter than other arterial grafts, and a thick, muscular wall that facilitates the construction of an anastomosis. However, early experience suggested that RA grafts were prone to spasm and functional occlusion, and their use was abandoned for many years. In the past decades, the advent of drug therapy to prevent graft spasm and the adoption of newer harvesting techniques revitalized the interest the use of radial artery. Recently several randomized trials has been conducted to prove the better graft patency over the saphenous vein (SV) and survival benefit was also observed as well. However, due to its unneglectable vulnerability to competitive flow, the recent American and European guidelines for coronary revascularization both limited the use of RA only in significantly stenosed vessels.

Fractional flow reserve (FFR) is the current gold standard to measure the physiological significance of coronary stenosis and the potential for competitive flow. The quantitative flow ratio (QFR) is a novel, intelligent, noninvasive method that enables efficient computation of the FFR from coronary angiography in good concordance with catheter-based FFR. QFR-guided percutaneous coronary intervention (PCI) has been used and showed the improved clinical outcomes in FAVOR III China trial (Comparison of Quantitative Flow Ratio-Guided and Angiography-Guided Percutaneous InterVention in Patients With cORonary Artery Disease).

The Impact of Preoperative Quantitative Flow Ratio on Radial-Artery Graft Outcome after Coronary Artery Bypass Grafting (ASRAB-QUARGO) study aims to investigate whether the preoperative QFR measurement is associated with RA graft patency 6 months after CABG, and to explore the best QFR cut-off value for guiding RA-CABG.

Methods:

Study design- The ASRAB-QUARGO is a single-centre, prospective, double-blind, observational sub-study of the ASRAB-pilot trial (NCT04310995). The study was registered and approved by the ethics committee in out institution. Informed consent was waived under permission from the ethics committee.

Outcome- The primary outcome is the association between preoperative QFR of target vessel and the RA graft outcome at 6 months after CABG. The secondary outcome is the association between preoperative QFR of target vessel and the RA graft outcome at 7 days after CABG.

Study procedures- The complete eligibility criteria for ASRAB-pilot trial is provided in the "eligibility" section. After successfully receiving primary isolated CABG, the patients from the ASRAB-pilot cohort with preoperative CAG images available for QFR analysis were enrolled in this study. QFR analysis was conducted in all vessels grafted based on preoperative CAG images. The images were sent to the core lab (CardHemo, Med-X Research Institute, Shanghai Jiao Tong University, Shanghai, China) for computation of the QFR. The analysis was performed by the experienced analysts using the AngioPlus system (Pulse Medical Imaging Technology, Shanghai, China) as described [11-15]. QFR results were recorded by the core lab and blinded to the patient and surgeon. Apart from the investigational anti-spastic drug from the ASRAB-pilot trial, optimized medical treatment was pursued according to the current American and European guidelines, including smoking cessation counselling and the administration of antiplatelet agents, beta blockers, lipid medications, and angiotensin-converting enzyme inhibitors.

Patients underwent follow-up coronary computer tomography angiography （CCTA）6 months after surgery. Angiographic evaluations were performed by two observers (one radiologist and one cardiac surgeon) blinded to the preoperative QFR values. In the case of ambiguity or disagreement between observers, additional CAG is conducted as possible for further confirmation. For sequential grafts, each segment between two adjacent anastomoses (graft-to-graft anastomosis not included) will be defined as an independent graft and evaluated independently. For composite grafts (eg. T or Y grafts), only RAs directly anastomosed to target vessel were considered as RA grafts. Angiographic patency was graded referring to the FitzGibbon classification: 4 Grade A for widely patent, Grade B for patent with flow limited, Grade S for string sign and Grade O for occluded. Grade B, O and S were considered as diseased. MACE was defined as a composite of all-cause death, nonfatal myocardial infarction, nonfatal stroke and unplanned coronary revascularization.

Sample size- Historical data from our center indicate that graft disease (Grade B, O & S) occurs in around 20% of grafts 6 months after CABG. We estimated an RA graft disease rate of 10% if QFR ≤ best cut-off value (0.50-0.55 assumed), and 30% if QFR > best cut-off valve (0.5-0.55 assumed). With a power of 0.80 at an alpha level of 0.05, 118 RA grafts would be required to detect a statistically significant difference between groups. Assuming a 10% dropout rate and an average of 1.2 anastomosis per patient, sample size was defined at 110 patients. Therefore, the cohort size of ASRAB-pilot study of 150 patients is deemed adequate.

Analytic design and statistical analysis- Continuous variables were reported as mean, standard deviation, median, interquartile, minimum or maximum. For discrete categorical data, statistical description was presented as count and percentage. Missing data was treated as random missing. Unless otherwise stated, missing data was not filled in in this study.

Considering the possible heterogeneity between the sample population and the actual population for application, 2000 resampling samples were constructed through bootstrapping, and the mean value of QFR cut-off of all samples was taken as the final QFR cut-off. The determination of QFR cut-off value for a single sample adopted the minimum p-value method, taking RA, ITA or SV graft disease at 6 months after operation as endpoint index.

Considering the observational nature of this study, the cohort grouped based on the QFR cut-off may had imbalance of important factors. Therefore, the multivariate regression model and propensity scoring method were used to correct the potential confounding factors to evaluate the difference of outcome indicators between groups after the QFR cut-off grouping. The correlation between QFR and visual estimation was analyzed by the Spearman rank-order correlation coefficient. The predictive value of QFR and visual estimation for graft disease was compared by analyzing their respective ROC curve and corresponding AUC. Taking the QFR and the visual estimation as important prediction variables, a multifactor prediction model was constructed. The prediction accuracy was evaluated and compared by AUC. The prediction model was presented as nomograms, and the calibration curve and decision analysis curve were constructed.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the ASRAB-pilot study.

Exclusion Criteria:

* Preoperative CAG not available for QFR analysis.

The inclusion and exclusion criteria of ASRAB-pilot study are attached:

Inclusion Criteria:

* Age≥18 years.
* Male or female patients.
* Have signed informed consent.
* Have successfully accepted the first RA-CABG surgery.

Exclusion Criteria:

* Previously experienced an allergy to active ingredients and/or excipients of experimental drugs.
* Hypotension (defined as systolic blood pressure < 90mmHg or diastolic blood pressure < 60mmHg) after surgery.
* Acute myocardial infarction, pulmonary congestion or cardiogenic shock after surgery.
* Concomitant medications with phosphodiesterase-5 inhibitors such as sildenafil, vardenafil, tadalafil, etc.
* Pathological sinus node syndrome, degree II or III atrioventricular block without cardiac pacemaker.
* Contraindications for coronary computed tomography angiography (CCTA) or coronary arteriography (CAG) examination, such as iodine allergy, etc. (note: patients with renal insufficiency or even end-stage renal disease whose hemodialysis can be tolerated by CCTA or CAG tests are eligible for inclusion).
* History or evidence of ongoing alcohol or drug abuse.
* Life expectancy < 1 year judged by investigators.
* Other inappropriate situations judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patients enrolled in the ASRAB-pilot trial, those who with available preoperative CAG images for QFR analysis, will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
6-month radial artery graft failure | 6 months after surgery
  Graft outcome will be evaluated by CCTA or CAG according to the Fitzgibbon classification criteria: Grade A, grade B, grade O and grade S (String Sign). Grade B, O and S are considered as graft failure.
7-day radial artery graft failure | 7 days after surgery
  Graft outcome will be evaluated by CCTA or CAG according to the Fitzgibbon classification criteria: Grade A, grade B, grade O and grade S (String Sign). Grade B, O and S are considered as graft failure.

SECONDARY OUTCOMES:
Major adverse cardiovascular event (MACE) | within 6 months after surgery
  MACE is defined as a composite of all-cause death, myocardial infarction, stroke and unplanned coronary revascularization. The first occurring MACE or its component, as well as the time of occurrence, is collected.
Myocardial infarction related to radial artery graft failure | within 6 months after surgery
  Defined as new wall motion abnormalities detected by echocardiogram, or new Q wave detected by electrocardiograph (ECG) in the region grafted with radial artery.
Unplanned coronary revascularization related to radial artery graft failure | within 6 months after surgery
  Subjects may receive unplanned revascularization to the territory originally grafted by radial artery graft, either by PCI or CABG. This is defined as an "unplanned coronary revascularization related to radial artery graft failure" event.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD, Principal Investigator — Ruijin Hospital; Yunpeng Zhu, MD, Study Director — Ruijin Hospital; Jiaxi Zhu, MD, Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):e652-735. doi: 10.1161/CIR.0b013e31823c074e. Epub 2011 Nov 7. No abstract available. PMID 22064599
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Lytle BW, Blackstone EH, Loop FD, Houghtaling PL, Arnold JH, Akhrass R, McCarthy PM, Cosgrove DM. Two internal thoracic artery grafts are better than one. J Thorac Cardiovasc Surg. 1999 May;117(5):855-72. doi: 10.1016/S0022-5223(99)70365-X. PMID 10220677
- [Background] Taggart DP, D'Amico R, Altman DG. Effect of arterial revascularisation on survival: a systematic review of studies comparing bilateral and single internal mammary arteries. Lancet. 2001 Sep 15;358(9285):870-5. doi: 10.1016/S0140-6736(01)06069-X. PMID 11567701
- [Background] Yi G, Shine B, Rehman SM, Altman DG, Taggart DP. Effect of bilateral internal mammary artery grafts on long-term survival: a meta-analysis approach. Circulation. 2014 Aug 12;130(7):539-45. doi: 10.1161/CIRCULATIONAHA.113.004255. Epub 2014 Jun 10. PMID 24916209
- [Background] Aldea GS, Bakaeen FG, Pal J, Fremes S, Head SJ, Sabik J, Rosengart T, Kappetein AP, Thourani VH, Firestone S, Mitchell JD; Society of Thoracic Surgeons. The Society of Thoracic Surgeons Clinical Practice Guidelines on Arterial Conduits for Coronary Artery Bypass Grafting. Ann Thorac Surg. 2016 Feb;101(2):801-9. doi: 10.1016/j.athoracsur.2015.09.100. Epub 2015 Dec 8. PMID 26680310
- [Background] Glineur D, Poncelet A, El Khoury G, D'hoore W, Astarci P, Zech F, Noirhomme P, Hanet C. Fractional flow reserve of pedicled internal thoracic artery and saphenous vein grafts 6 months after bypass surgery. Eur J Cardiothorac Surg. 2007 Mar;31(3):376-81. doi: 10.1016/j.ejcts.2006.11.023. Epub 2006 Dec 14. PMID 17174100
- [Background] Glineur D, Hanet C. Competitive flow in coronary bypass surgery: is it a problem? Curr Opin Cardiol. 2012 Nov;27(6):620-8. doi: 10.1097/HCO.0b013e3283583000. PMID 23075821
- [Background] Glineur D, D'hoore W, El Khoury G, Sondji S, Kalscheuer G, Funken JC, Rubay J, Poncelet A, Astarci P, Verhelst R, Noirhomme P, Hanet C. Angiographic predictors of 6-month patency of bypass grafts implanted to the right coronary artery a prospective randomized comparison of gastroepiploic artery and saphenous vein grafts. J Am Coll Cardiol. 2008 Jan 15;51(2):120-5. doi: 10.1016/j.jacc.2007.09.030. PMID 18191734
- [Background] Glineur D, Hanet C, D'hoore W, Poncelet A, De Kerchove L, Etienne PY, Noirhomme P, El Khoury G. Causes of non-functioning right internal mammary used in a Y-graft configuration: insight from a 6-month systematic angiographic trial. Eur J Cardiothorac Surg. 2009 Jul;36(1):129-35; discussion 135-6. doi: 10.1016/j.ejcts.2009.02.041. Epub 2009 Apr 15. PMID 19372044
- [Background] Sabik JF 3rd, Lytle BW, Blackstone EH, Khan M, Houghtaling PL, Cosgrove DM. Does competitive flow reduce internal thoracic artery graft patency? Ann Thorac Surg. 2003 Nov;76(5):1490-6; discussion 1497. doi: 10.1016/s0003-4975(03)01022-1. PMID 14602274
- [Background] White CW, Wright CB, Doty DB, Hiratza LF, Eastham CL, Harrison DG, Marcus ML. Does visual interpretation of the coronary arteriogram predict the physiologic importance of a coronary stenosis? N Engl J Med. 1984 Mar 29;310(13):819-24. doi: 10.1056/NEJM198403293101304. PMID 6700670
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Background] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Tu S, Westra J, Adjedj J, Ding D, Liang F, Xu B, Holm NR, Reiber JHC, Wijns W. Fractional flow reserve in clinical practice: from wire-based invasive measurement to image-based computation. Eur Heart J. 2020 Sep 7;41(34):3271-3279. doi: 10.1093/eurheartj/ehz918. PMID 31886479
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Background] Glineur D, Grau JB, Etienne PY, Benedetto U, Fortier JH, Papadatos S, Laruelle C, Pieters D, El Khoury E, Blouard P, Timmermans P, Ruel M, Chong AY, So D, Chan V, Rubens F, Gaudino MF. Impact of preoperative fractional flow reserve on arterial bypass graft anastomotic function: the IMPAG trial. Eur Heart J. 2019 Aug 1;40(29):2421-2428. doi: 10.1093/eurheartj/ehz329. PMID 31155673
- [Background] Glineur D, Rahouma M, Grau JB, Etienne PY, Fortier JH, Papadatos S, Laruelle C, Pieters D, El Khoury E, Gaudino M. FFR Cutoff by Arterial Graft Configuration and Location: IMPAG Trial Insights. JACC Cardiovasc Interv. 2020 Jan 13;13(1):143-144. doi: 10.1016/j.jcin.2019.08.013. No abstract available. PMID 31918937